CLINICAL TRIAL: NCT01136187
Title: ST Elevation Myocardial Infarction Treated by RADIAL or Femoral Approach - Randomized Multicenter Study Comparing Radial Versus Femoral Approach in Primary PCI. The STEMI-RADIAL Trial.
Brief Title: Trial Comparing Radial and Femoral Approach in Primary Percutaneous Coronary Intervention (PCI)
Acronym: STEMI-RADIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: University Hospital Pilsen (Other); Regional Hospital Liberec (Other); University Hospital Hradec Kralove (Other); Na Homolce Hospital (Other)
Responsible Party: Principal Investigator, Ivo Bernat, MD, PhD, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STEMI-RADIAL 16-9-2009
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Myocardial infarction; Primary percutaneous coronary intervention; Radial; Bleeding
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction; Hemorrhage

ARMS (2):
- Radial approach (Experimental): Primary percutaneous coronary intervention from the radial approach
  Interventions: Procedure: Access site in primary PCI
- Femoral approach (Active Comparator): Primary percutaneous coronary intervention from the femoral approach
  Interventions: Procedure: Access site in primary PCI

INTERVENTIONS:
Procedure: Access site in primary PCI

SUMMARY:
Percutaneous coronary interventions (PCIs) from the femoral approach have more bleeding complications related to access site in comparison to the radial approach in patients with acute coronary syndrome (ACS). Major bleeding and access site complications have an important role in results of PCI for ACS and lead to higher morbidity and mortality. Primary PCIs in ST elevation myocardial infarction (STEMI) are associated with more aggressive antithrombotic treatment than in elective or semi-urgent interventions. Currently, both radial and femoral approaches are routinely used for primary PCI in STEMI. However, only non-randomized studies and registries or small randomized single center studies comparing both approaches in primary PCI have been published until now. The aim of STEMI-RADIAL trial is to evaluate potential reduction of bleeding complications in the radial approach primary PCI compared to femoral approach in randomized, multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Admission for STEMI less than 12 hours after onset of symptoms

  1. Patients have typical chest pain for at least 20 minutes and have ECG changes typical for STEMI (ST elevation ≥ 2 mm in two continuous precordial leads or ST elevations ≥ 1 mm in two limb leads or new left bundle branch block) or ECG changes compatible with true posterior MI.
  2. Patients are planned to be treated with primary PCI
* Ability to sign written informed consent

Exclusion Criteria:

* Killip IV class or unconsciousness
* Patient disagreement
* Prior aortobifemoral bypass
* Absence of both radial or femoral artery pulsation
* Participation in another clinical trial randomizing ACS patients using antithrombotic drug.
* Negative Allen's test or Barbeau test type D
* Treatment with oral anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of bleeding or entry site complications | 30 days

SECONDARY OUTCOMES:
Occurence of major adverse cardiovascular events
Primary access site failure - conversion to another access
Angiographical procedural success
Contrast media consumption
Procedural and fluoroscopic times
Duration of hospital / ICU stay
TVR/TLR + any new hospitalization

CONTACTS AND LOCATIONS:
Locations (4):
- Czechia (4):
  - University Hospital Hradec Kralove, Hradec Králové
  - Regional Hospital Liberec, Liberec
  - University Hospital Pilsen, Pilsen
  - Na Homolce Hospital, Prague

REFERENCES:
- [Derived] Bernat I, Horak D, Stasek J, Mates M, Pesek J, Ostadal P, Hrabos V, Dusek J, Koza J, Sembera Z, Brtko M, Aschermann O, Smid M, Polansky P, Al Mawiri A, Vojacek J, Bis J, Costerousse O, Bertrand OF, Rokyta R. ST-segment elevation myocardial infarction treated by radial or femoral approach in a multicenter randomized clinical trial: the STEMI-RADIAL trial. J Am Coll Cardiol. 2014 Mar 18;63(10):964-72. doi: 10.1016/j.jacc.2013.08.1651. Epub 2013 Nov 21. PMID 24211309